CLINICAL TRIAL: NCT03187860
Title: Demonstration of the Diagnostic Character of the Rheology of Mucus
Brief Title: Ciliation and Mucus Rheology Parameters Determined Via Air-liquid-interface Cell Cultures in Non-smoking, Smoking, COPD and Asthmatic Patients
Acronym: RhéMuc
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusions was stopped at 30 patients. Investigators did not wish to extend inclusions.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL18_0222
Record Dates: First submitted 2017-06-12; First posted 2017-06-15 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma; Smoking
Keywords: Bronchial epithelial cell; mucus; Air Liquid Interface
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-smoking controls (Experimental): Subjects in this group have never smoked and have no known lung disorders.
  Intervention: Bronchial Biopsy + ALI culture (Air Liquid Interface)
  Interventions: Procedure: Bronchial Biopsy; Other: ALI culture
- Smokers without COPD (Experimental): Subjects in this group are smokers or former smokers who do not have signs of obstructive disease (no chronic obstructive pulmonary disease (COPD))
  Intervention: Bronchial Biopsy + ALI culture
  Interventions: Procedure: Bronchial Biopsy; Other: ALI culture
- Smokers with COPD (Experimental): Subjects in this group are smokers or former smokers who have COPD
  Intervention: Bronchial Biopsy + ALI culture
  Interventions: Procedure: Bronchial Biopsy; Other: ALI culture
- Severe asthma (Experimental): Subjects in this group are non-smokers or former (light) smokers who have severe asthma.
  Intervention: Bronchial Biopsy + ALI culture
  Interventions: Procedure: Bronchial Biopsy; Other: ALI culture

INTERVENTIONS:
Procedure: Bronchial Biopsy — Bronchial biopsies will be performed on all subjects.
Other: ALI culture — Air-liquid-interface cell cultures will be derived from bronchial biopsy specimens. We are expecting several replicate cell lines from each biopsy specimen.

SUMMARY:
This is a prospective study comparing 4 groups: (1) non-smoking controls, (2) smokers without chronic obstructive pulmonary disease (COPD), (3) smokers with COPD, (4) severe asthma.

Bronchial biopsy specimens from each subject will be obtained to produce air-liquid-interface cell cultures. These will then be used to make observations concerning cilia and mucus rheology.

This is a first pilot study. The working hypothesis is that the largest group differences will be found for cilia densities; the latter metric was thus chosen as a primary criterion.

ELIGIBILITY:
Inclusion criteria for non smoking controls:

* The subject has given free and informed consent and signed the consent form
* The subject is affiliated with or beneficiary of a medical insurance program
* The subject has never smoked
* No obstructive breathing disorder (forced expiratory volume at one second (FEV1) >70% of predicted value; the ratio of FEV1 to forced vital capacity (FEV1/FVC) is > 0.7)
* No known respiratory disease

Inclusion criteria for smokers without COPD:

* The subject has given free and informed consent and signed the consent form
* The subject is affiliated with or beneficiary of a medical insurance program
* Smoker or former smoker (>= 30 pack years)
* No obstructive breathing disorder (forced expiratory volume at one second (FEV1) >70% of predicted value; the ratio of FEV1 to forced vital capacity (FEV1/FVC) is > 0.7)

Inclusion criteria for smokers with COPD:

* The subject has given free and informed consent and signed the consent form
* The subject is affiliated with or beneficiary of a medical insurance program
* Smoker or former smoker (>= 30 pack years)
* Subject presenting with COPD: FEV1/FVC < 0.7 (based on spirometry values in the medical file and performed in the 3 months prior to inclusion)
* The subject requires bronchial fibroscopy (decision made by pneumologist)
* COPD of grade "2" or "3" according to GOLD criteria (Global Initiative for Chronic Obstructive Lung Disease)

Inclusion criteria for subjects with severe asthma:

* The subject has given free and informed consent and signed the consent form
* The subject is affiliated with or beneficiary of a medical insurance program
* Non-smoker or former smoker (<10 pack years)
* Subject presenting with severe asthma: FEV1/FVC >= 0.7 and FEV1 < 80%
* The subjects requires bronchial fibroscopy (decision made by pneumologist)

Exclusion criteria:

* The subject has an extensive neoplastic disease
* The subject has another active lung disease (tuberculosis, pulmonary interstitium disease, active or recent pulmonary infection)
* The subject has had a recent psychiatric disorder (within one year prior to inclusion and documented by a specialist consultation)
* Emergency situations (object extractions...)
* Subject consuming illicit drugs or alcohol
* The subject is in an exclusion period determined by a previous study
* The subject is under judicial protection, or is an adult under any kind of guardianship
* It is impossible to correctly inform the patient
* The subject cannot fluently read French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
Surface density of active cilia | Day 0 + approximately 2 months of cell culture time
  Surface density of active cilia

SECONDARY OUTCOMES:
Cilia beating frequency | Day 0 + approximately 2 months of cell culture time
  The frequency at which cilia beat.
Mucus viscosity | Day 0 + approximately 2 months of cell culture time
  The viscosity of mucus produced by cell cultures.
Mucus elasticity | Day 0 + approximately 2 months of cell culture time
  The elasticity of mucus produced by cell cultures.
Cilia beat orientation | Day 0 + approximately 2 months of cell culture time
  The direction in which cilia beat

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sophie Gamez, MD, Study Director — Montpellier University Hospitals
Locations (1):
- CHU Montpellier, Montpellier, France